CLINICAL TRIAL: NCT02520115
Title: Study of Serum Measured Folate Receptor and Its Induction as a Biomarker in the Diagnosis and Surveillance of Ovarian Carcinoma
Brief Title: Folate Receptor in Diagnosing Ovarian Cancer Using Serum Samples From Patients With Newly Diagnosed Pelvic Mass or Previously Diagnosed Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ira Winer, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-024; NCI-2015-01039 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1504013983; 2015-024 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2015-07-30; First posted 2015-08-11 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Adnexal Mass; Borderline Ovarian Epithelial Tumor; Ovarian Clear Cell Tumor; Ovarian Endometrioid Tumor; Ovarian Neoplasm; Ovarian Serous Tumor; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (induction) (Experimental): Patients receive valproic acid PO BID on days -7 to -3 and QD on day -2 and dexamethasone PO QD on days -5 and -2 and BID on days -4 and -3. Patients undergo collection of serum and tissue samples for analysis via PCR and IHC at baseline, time of surgery, and 7-14 days after surgery.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Valproic Acid
- Arm II (surveillance and recurrence) (Experimental): Patients receive valproic acid PO BID on days -7 to -3 and QD on day -2 and dexamethasone PO QD on days -5 and -2 and BID on days -4 and -3. Patients undergo collection of serum samples for analysis via PCR and IHC at the time of clinically suspected recurrence, 2 days after completion of induction, and 7-14 days after induction.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Valproic Acid

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Analysis of serum and tissue samples
Drug: Valproic Acid — Given PO
  Other Names: Depakene; Stavzor; Valproate

SUMMARY:
This pilot research trial studies folate receptor in diagnosing ovarian cancer using serum samples from patients with a newly diagnosed pelvic mass or previously diagnosed ovarian cancer. Studying samples of serum from patients with ovarian cancer in the laboratory may help understand the use of folate receptor induction as a clinical tool in initial diagnosis, surveillance, and recurrence.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the pre- and post-induction correlation between soluble folate receptor and tumor-based receptor levels as a marker of malignancy in patients with newly diagnosed adnexal masses. (Arm I) II. To evaluate the ability to induce serum folate receptor (FR) with dexamethasone (Dex) and valproic acid (VPA) treatment in patients with newly diagnosed adnexal masses. (Arm I) III. To evaluate the use of the serum soluble FR as a marker for earlier detection of recurrent disease. (Arm II) IV. To evaluate the ability to induce FR with Dex and VPA in the setting of recurrent disease. (Arm II)

SECONDARY OBJECTIVES:

I. To evaluate the expression of FR in primary versus (vs.) metastatic tumor sites in patients with ovarian malignancy undergoing Dex and VPA induction and correlate expression with other markers associated with malignancy (marker of proliferation Ki-67 [Ki67], cancer antigen [CA]-125, etc.).

II. To analyze the correlation between gluco-corticoid receptor (GR) levels and serum FR induction efficacy.

III. To examine global, downstream targets of GR and FR induction in patient samples undergoing treatment with Dex and VPA.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (INDUCTION): Patients receive valproic acid orally (PO) twice daily (BID) on days -7 to -3 and once daily (QD) on day -2 and dexamethasone PO QD on days -5 and -2 and BID on days -4 and -3. Patients undergo collection of serum and tissue samples for analysis via polymerase chain reaction (PCR) and immunohistochemistry (IHC) at baseline, time of surgery, and 7-14 days after surgery.

ARM II (SURVEILLANCE AND RECURRENCE): Patients receive valproic acid PO BID on days -7 to -3 and QD on day -2 and dexamethasone PO QD on days -5 and -2 and BID on days -4 and -3. Patients undergo collection of serum and tissue samples for analysis via PCR and IHC at the time of clinically suspected recurrence, 2 days after completion of induction, and 7-14 days after induction.

ELIGIBILITY:
Inclusion Criteria:

* For study Arm 1, female subjects of childbearing potential or less than 2 years postmenopausal agree to use an acceptable form of contraception from the time of signing informed consent until 30 days after study completion unless total hysterectomy performed at the time of original operation
* Able to provide informed consent
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
* Study Arm 1: primary diagnosis of a pelvic or adnexal mass of presumed gynecologic origin who is scheduled for operative resection
* Study Arm 2: previously diagnosed with a non-mucinous epithelial ovarian carcinoma (including serous, clear cell, and endometrioid histologies as well as borderline ovarian tumors) currently undergoing routine surveillance for recurrence, having been diagnosed with recurrence but prior to initiation of chemotherapy. . Patients from Study Arm 1 will automatically be included in Study Arm 2 as well unless they withdraw consent. Finally, patients who have been diagnosed with an ovarian cancer of acceptable histology but not yet initiated adjuvant chemotherapy are eligible for Study Arm 2.

Exclusion Criteria:

* Known sarcomatous histologies
* Current usage of VPA or Dex, if patient has been on these medications in the past but is not currently taking them she is still a candidate for the study. Prior use must be greater than one month for VPA. There is no "wash out" period required for DEX.
* Any contraindication to dexamethasone or valproic acid such as known allergies or sensitivity
* Unable to give informed consent
* Pregnancy
* Greater than 3 x the upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST)
* Greater than 3 x the ULN for total bilirubin (except for known cases of Gilbert's syndrome, where the levels of conjugated bilirubin must be less than 3 x the ULN)
* Greater than 1.5 x the ULN for blood urea nitrogen (BUN)
* Greater than 1.5 x the ULN for creatinine
* Chronic or acute pancreatitis as evidenced by clinical or pathologic diagnosis
* Significant acute or chronic medical, neurologic, or psychiatric illness in the subject that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study
* For study Arm 2, patients that are currently undergoing chemotherapy for recurrence; maintenance chemotherapy is not considered an exclusion criteria. Additionally, as noted above if a patient has not yet begun chemotherapy for recurrence or adjuvant chemotherapy for initial diagnosis they are still a candidate to be enrolled on this Study arm.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2018-09 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Arm I: To evaluate the ability to increase serum Folate Receptor (FR) levels in patients with newly diagnosed adnexal masses or ovarian cancer utilizing Dexamethasone (DEX) and Valproic Acid (VA). | Up to 14 days after induction
  FR will be measured in the serum of patients utilizing a standardized tritiated folate/charcoal binding assay pre- and post-drug administration. This will be measured to the femto-molar level. Two sided t-tests will be utilized as a baseline statistical analysis to determine the efficacy of induction in this setting.
Arm I: To evaluate the utility of serum FR to distinguish between patients with benign masses or malignancy. | Up to 14 days after surgery
  Folate receptor levels in patients with benign and malignant conditions will be compared utilizing receiver operator curves for both pre- and post-induction levels to determine if soluble folate receptor can be utilized as a tumor marker in newly diagnosed adnexal masses and/or ovarian cancer. Both two-sided t tests and ROC curve analysis will be utilized in this portion of the analysis.
Arm II: To evaluate the use of the serum soluble FR as a marker for earlier detection of recurrent disease. | Up to 14 days after induction
  Patients are to be followed during surveillance period for a history of know ovarian carcinoma with serum FR in addition to CA-125. FR will again be measured in the serum of patients utilizing a standardized tritiated folate/charcoal binding assay. This will be measured to the femto-molar level. ROC curve analysis will be performed to evaluate the efficacy of baseline Folate Receptor in early detection of relapse and compared to standard tumor markers such as CA-125.
Arm II: To evaluate the ability to increase serum FR levels with DEX and VA in the setting of recurrent disease. | Up to 14 days after surgery
  If recurrence is suspected, this portion of Arm 2 is meant to determine if serum levels of FR can be artificially increased in the recurrent setting utilizing DEX and VA above baseline recurrent levels. FR will be measured in the serum of patients utilizing a standardized tritiated folate/charcoal binding assay pre- and post-drug administration. This will be measured to the femto-molar level. Two side t-tests will be utilized to determine the efficacy of induction in this setting.

SECONDARY OUTCOMES:
Arm I: To evaluate expression of FR via immunohistochemistry in primary vs. metastatic tumor sites in patients with ovarian malignancy undergoing DEX & VA induction and determine if this correlates with other known markers associated with malignancy. | Up to day 14
  Two sided independent t-tests will be performed to compare the expression of FR in primary vs metastatic tumor sites. Pearson's correlation coefficients will be calculated to evaluate the associations between serum FR and existing markers such as Ki67 and CA-125.
Arm I: To examine downstream targets of GR and FR induction in patient samples undergoing treatment with DEX and VA via global mRNA analysis and proteomic modalities. | Up to day 14
  Achieved by utilizing such techniques (but not limited to) as transcriptome analysis and whole genome Chip analysis.
Arm I: To analyze the correlation between GR level as noted by immunohistochemistry and serum FR induction efficacy with DEX and VA. | Up to day 14
  Pearson's correlation coefficients will be calculated to evaluate the associations between serum Folate receptor levels and tissue based glucocorticoid receptors.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Winer, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Karmanos Cancer Institute at McLaren Bay Region, Bay City, Bay City, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan